CLINICAL TRIAL: NCT02754414
Title: Cold Apheresis Platelets in PAS
Acronym: CAPP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bloodworks (Other)
Responsible Party: Principal Investigator, Moritz Stolla, MD, Director, Platelet Transfusion Research, Bloodworks
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016 - 01; CAPI (Other: BloodworksNW)
Record Dates: First submitted 2016-04-07; First posted 2016-04-28 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Platelet Transfusion
Keywords: platelets; transfusion; cold storage; apheresis
MeSH Terms: interventions — In Vitro Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Volunteers (Experimental): Autologous, cold stored, PAS/plasma suspended platelets stored for various periods (3 to 20 days).
  Interventions: Procedure: Apheresis platelet collection; Other: Refrigerated storage of apheresis platelets in PAS/plasma; Radiation: Infusion of aliquot of autologous radiolabeled platelets; Other: In vitro tests

INTERVENTIONS:
Procedure: Apheresis platelet collection — A single apheresis platelet unit will be collected from a healthy adult volunteer subject using the Trima Accel® Automated Blood Collection System. Concurrent plasma will be collected.
Other: Refrigerated storage of apheresis platelets in PAS/plasma — The apheresis platelet unit will be stored, without agitation, at 4°C, for up to 20 days.
Radiation: Infusion of aliquot of autologous radiolabeled platelets — Fresh and stored aliquots will be labeled with Indium-111. We are administering ≤30 microcuries in both infusions for a total dose of 0.8 mSv.
Other: In vitro tests — Tests to evaluate platelet function will be performed on the platelet unit on day of collection and end of storage

SUMMARY:
This is a platelet transfusion study. The purpose of this study is to measure the life span and quality of platelets stored in a refrigerator. Participants will give platelets by apheresis. Platelets will be stored for 3 -20 days. A small portion of the subject's own stored platelets will be tagged with a radioactive isotope and infused back into the participant. This will enable us to track how many transfused platelets survive after storage in the refrigerator.

DETAILED DESCRIPTION:
A single hyperconcentrated apheresis platelet unit will be collected from a healthy adult volunteer subject using the Trima Accel® Automated Blood Collection System. Concurrent plasma will be collected. The platelet unit will be stored, not-agitated, for up to 20 days at 4°C in a suspension of 35% plasma and 65% PAS (Platelet Additive Solution).

At the end of the storage period, the subject will return to receive an 111Indium Oxine (Indium 111, In-111) radiolabeled aliquot of their 4°C stored platelets. Follow-up samples from the subject will be collected approximately 2 hours post-infusion and on Days 1 (2X), 2 (2X), and 3 to calculate recovery and survival of the subject's 4°C stored platelets. The Day 1 and Day 2 the sample draws will be 2 - 10 hours apart.

In addition to radiolabeled platelet recovery and survival measurements, various in vitro assays will be performed on the day of collection at the end of 4°C storage.

One week after the infusion of the radiolabeled aliquot, the subject will return to receive a second radiolabeled aliquot of fresh platelets. To facilitate this, on the morning of the second infusion, the subject will return for collection of a 43 mL blood sample. The blood will be processed to obtain a fresh sample of the subject's platelets to serve as a control comparator. The platelets will be radiolabeled with In-111. The subject will return later in the day for infusion of the radiolabeled fresh 'control' comparator aliquot. Follow-up blood samples will be drawn at ~2 hours after the infusion on Day 0 and then on Days 1, 2, 3, 4 or 5, and 6 or 7 day post infusion to calculate recovery and survival of the subject's fresh vs. stored platelets.

ELIGIBILITY:
Inclusion Criteria:

* Weight: ≥ 110 pounds
* Platelet count: ≥ 150X10^3/mL
* Hematocrit: 38% for females, 39% for males, but not >55%
* Temperature: ≤ 99.5 F
* Resting blood pressure: systolic ≤180 mmHg; diastolic ≤ 100 mmHg
* Resting heart rate: 40 to 100 beats per minute
* Subjects must be: at least 18 years old, of either sex
* Subjects must be able to read, understand and sign the informed consent document and commit to the study follow-up schedule. The ability to read and speak English is required for participation.
* Subjects must have good veins for apheresis platelet collection and drawing blood samples.
* Subjects of child-bearing potential (either male or female) must agree to use an effective method of contraception during the course of the study. The following methods of contraception are be considered effective; abstinence, intrauterine contraception devices, hormonal methods, barrier methods or history of sterilization.

Exclusion Criteria:

Healthy subjects will be excluded from the study for any of the following reasons:

* Unable to achieve target platelet yield of 3.0 X 1011/unit per Trima Accel (apheresis machine) configuration parameters.
* Ever received radiation therapy.
* Already participated in 4 research studies involving radioisotopes within the contemporaneous calendar-year.
* Taken aspirin, non-steroidal anti-inflammatory, or other platelet affecting drugs within 72 hours of collection or infusion. Subjects who have ever been prescribed anti-platelet medications (e.g. clopidogrel) will be excluded from study participation regardless of the interval to their last dose.
* Currently pregnant or nursing as assessed during interview. A urine pregnancy test prior to radioisotope infusion is required for women of childbearing potential.
* Unable to comply with the protocol in the opinion of the investigator.
* Donated granulocytes within the last 2 days.
* Donated whole blood within the last 7 days.
* Donated platelets or plasma within the last 28 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Maximal storage time with acceptable recovery and survival (as defined below) | up to 20 days storage at 4°C
  Tables of recovery and survival summary statistics will display values by group from fresh and stored platelets. Recovery and survival of stored platelets as percentage of corresponding fresh platelets will be plotted against days stored. Regression methods will be used to determine if there is evidence of any trend in the mean storage or recovery of 4°C stored platelets with respect to storage time as a percentage of each subject's fresh platelet results. Histograms of recovery and survival as percentage of 4°C stored platelet measurements will be plotted, and corresponding confidence intervals will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Bloodworks Northwest (formerly Puget Sound Blood Center), Seattle, Washington, United States